CLINICAL TRIAL: NCT02971644
Title: Cobalt Alloy Pedicle Screw Implantation for Severe Kyphosis Deformity in Spinal Tuberculosis: a Selfcontrolled Trial
Brief Title: Cobalt Alloy Pedicle Screw Implantation for Severe Kyphosis Deformity in Spinal Tuberculosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Affiliated Hospital of Hebei University (Other)
Responsible Party: Principal Investigator, Yu Hou, Associate Chief Physician, Affiliated Hospital of Hebei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HebeiU_001
Record Dates: First submitted 2016-11-14; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Spinal Tuberculosis
MeSH Terms: conditions — Tuberculosis, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cobalt alloy pedicle screw implantation (Experimental): The spinal tuberculosis patients with severe kyphosis deformity who will undergo cobalt alloy pedicle screw implantation.
  Interventions: Device: cobalt alloy pedicle screw implantation

INTERVENTIONS:
Device: cobalt alloy pedicle screw implantation — The patients with severe kyphosis deformity undergo cobalt alloy pedicle screw implantation.

SUMMARY:
To investigate whether implantation of cobalt alloy pedicle screws is effective in treating severe kyphosis deformity in spinal tuberculosis, and to determine the factors that are likely to have influenced the curative effects.

DETAILED DESCRIPTION:
History and current related studies The incidence of spinal tuberculosis has continually increased in recent years; this disease commonly occurs in the lumbar spine, lumbar vertebrae, thoracic vertebrae, and cervical vertebrae. The majority of spinal tuberculosis patients present with kyphosis deformity in corresponding segments. In spinal tuberculosis patients with severe kyphotic deformity, the key to successful treatment is the individual patient's response to tuberculosis drugs and the implementation of rational fixation approaches at an appropriate time; good curative effects have been shown using anterior or posterior fixation, followed by posterior debridement and bone graft fusion.

Surgery via the posterior or anterior approach will be respectively performed in 16 of 32 patients with tuberculosis of the lumbar spine. The spinal cord function of these 32 patients has been assessed as Frankel grade C (n = 7), D (n = 14) and E (n = 11). The primary outcome measure of this study will be the Cobb angle at the thoracic spine segments preoperatively versus 2 years postoperatively, which will be used to evaluate the postoperative change in the thoracic spine curvature. The primary causes of poor healing or recurrence of spinal tuberculosis at the thoracic and lumbar segments are reportedly improper surgical timing, poor debridement, improper selection of internal fixation methods, poor selection of bone graft material or grafting position, irregular anti-tuberculosis bacilli chemotherapy, drug tolerance, poor braking, and not using a brace after surgery. However, the factors that influence curative effects require further investigation.

Pedicle screws are commonly used to repair spine fracture, and therefore they should have good biocompatibility. Cobalt alloy reportedly exhibits good anti-bending and anti-compressive strength, strong impact toughness, good elastic modulus, small thermal expansion coefficient, and good compatibility with the human body. However, few studies have investigated the use of cobalt alloy pedicle screws for treatment of severe kyphosis deformity in spinal tuberculosis.

Adverse events The investigators will record adverse events, including vertebral body displacement, thoracic and lumbar back muscle injury, nonspecific low back pain, and screw pull out or loosening. If severe adverse events occur, investigators will report details, including the data of occurrence and measures taken to treat the adverse events, to the principle investigator and the institutional review board within 24 hours.

Data collection, management, analysis and open-access Data collection: Case report forms with demographic data, disease diagnosis, accompanying diseases, drug allergy history, and adverse events will be collected, processed using Epidata software (Epidata Association, Odense, Denmark), collated, and then recorded electronically by data managers using a double-data entry strategy.

Data management: The locked electronic database will be accessible and locked only by the project manager, and will not be altered. All data regarding this trial will be preserved by the Affiliated Hospital of Hebei University, China.

Data analysis: The electronic database will be statistically analyzed by a professional statistician who will create an outcome analysis report that will be submitted to the lead researchers. An independent data monitoring committee will supervise the mange the trial data, ensuring a scientific and stringent trial to yield accurate and complete data.

Data open access: Anonymized trial data will be published at www.figshare.com.

Statistical analysis Statistical analysis will be performed using SPSS 19.0 software, and will follow the intention-to-treat principle. Normally distributed measurement data will be expressed as mean ± standard deviation, and minimums and maximums. Non-normally distributed measurement data will be expressed as lower quartile (q1), and median and upper quartile (q3). The Wilcoxon matched pairs test will be performed for comparison of the Cobb angle preoperatively versus 2 years postoperatively. The Wilcoxon signed-rank test will be performed for comparison of pre- and post-operative Frankel grade, and McNemar's chi-squared test will be used to analyze the incidence of adverse reactions. Multiple logistic regression analysis will be performed to analyze the factors that influence curative effects, with calculation of regression coefficients, odd ratios and 95% confidence interval. The significance level will be α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of spinal tuberculosis
* Diagnosed with spinal tuberculosis via X-ray or MRI
* Spinal tuberculosis patients with severe kyphosis deformity at the thoracic and lumbar segments and a spinal Cobb angle ≥ 90° complicated by spinal cord compression or neurological dysfunction, spinal stability destruction and paravertebral abscess
* Frankel grade C, D, or E
* Age 24-67 years
* Provision of complete medical data
* Receiving anti-tuberculosis medication for 3 weeks

Exclusion Criteria:

* Inability to tolerate surgery
* Other concomitant spine diseases
* Unable or unwilling to participate in this clinical trial

Ages: 24 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Cobb angle | 2 years postoperatively
  A greater Cobb angle indicates more severe kyphosis deformity.

SECONDARY OUTCOMES:
X-ray image | baseline and 2 years postoperatively
  Anterior-posterior X-ray images of the scoliotic spine will be taken using a digital X-ray scanner.
Frankel Grade | baseline and 2 years postoperatively
  To evaluate the recovery of spinal cord function. The Frankel Grade classification is used to assess the severity of spinal cord injury.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hou, Master, Principal Investigator — Affiliated Hospital of Hebei University

IPD SHARING:
Plan to Share IPD: Undecided